CLINICAL TRIAL: NCT05410197
Title: Envofolimab and Lenvatinib in Combination With Gemcitabine Plus Cisplatin for Patients With Advanced Biliary Tract Cancer as First-Line Treatment: A Single-arm, Open-label, Phase II Study
Brief Title: Envofolimab and Lenvatinib Combined With Gemcitabine Plus Cisplatin for Advanced BTC as First-Line Treatment(ENLIGHTEN)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Ming Kuang, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BTC2022
Record Dates: First submitted 2022-06-04; First posted 2022-06-08 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Advanced Biliary Tract Cancer
Keywords: Advanced Biliary Tract Cancer; First-Line Treatment
MeSH Terms: interventions — lenvatinib; Gemcitabine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Envofolimab + Lenvatinib + Gemcitabine + Cisplatin (Experimental): Single-arm trial whereby all consented, enrolled, eligible patients receive Envofolimab, Lenvatinib, Gemcitabine and Cisplatin
  Interventions: Drug: Envofolimab; Drug: Lenvatinib; Drug: Gemcitabine; Drug: Cisplatin

INTERVENTIONS:
Drug: Envofolimab — 400mg by subcutaneous injection every 3 weeks
Drug: Lenvatinib — 8 mg orally once a day
Drug: Gemcitabine — 1000mg/m2 by intravenous infusions on day 1 and 8 every 3 weeks for up to 24 weeks
Drug: Cisplatin — 25mg/m2 by intravenous infusions on day 1 and 8 every 3 weeks for up to 24 weeks

SUMMARY:
This is a phase 2, single-arm, open label study. The purpose is to investigate both the efficacy and safety of Envofolimab and Lenvatinib in combination with Gemcitabine plus Cisplatin for treatment of advanced biliary tract cancer as first-line treatment.

DETAILED DESCRIPTION:
The trial will recruit 43 patients. At the first step, 10 patients will be recruited. Only when at least 4 patients achieve objective response will the trial enter the second step and continue to recruit other patients. After being enrolled, all patients giving written informed consent will receive treatment until progression of disease, unacceptable toxicity or death. The tumor response evaluation will be conducted on a regular basis until progression of disease. Long-term survival follow up will be conducted as well.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent obtained from the patient prior to treatment.
2. Age > 18 years at the time of study entry.
3. Pathologically confirmed advanced biliary tract cancer, not having received systemic therapy.
4. Measurable or evaluable lesions according to RECIST v1.1 criteria.
5. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1.
6. Life expectancy ≥ 12 weeks.
7. Adequate hematologic (absolute neutrophil count ≥ 1,500/μL, platelets count ≥ 100,000/μL, hemoglobin ≥ 9.0 g/dL), renal (serum creatinine ≤ 1.5 × upper limit of normal (ULN) or creatinine clearance ≥ 50 mL/min (Cockcroft-Gault), urinary protein < 2+ or ≤ 1g/24h) and hepatic function (total serum bilirubin ≤ 1.5 ×ULN, serum aspartate aminotransferase (AST) and serum alanine aminotransferase (ALT) ≤ 2.5 × ULN).
8. Normal coagulation function (INR ≤ 1.5 × ULN, APTT ≤ 1.5 × ULN, PT ≤ 1.5 × ULN), without active bleeding or thrombotic diseases.
9. Willingness and ability to comply with the protocol.

Exclusion Criteria:

1. Diagnosis of any second malignancy, except for adequately treated basal cell skin cancer or in situ carcinoma of the cervix uteri.
2. Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients.
3. Previous treatment with Chinese herbal medicine or immunomodulators within 2 weeks, or radiotherapy treatment within 4 weeks prior to the first dose of administration.
4. Abnormal thyroid function.
5. Uncontrolled hypertension.
6. Uncontrolled cardiac disease, including but not limited to heart failure (NYHA class II-IV), unstable angina pectoris, myocardial infarction within 1 year or cardiac arrhythmia.
7. Active or prior documented autoimmune or inflammatory disorders.
8. Any immunosuppressants or systemic steroid therapy (> 10 mg daily dose of prednisone or equivalent) within 2 weeks prior to enrollment.
9. Central nervous system metastases.
10. Active infection or unknown fever(>38.5℃) prior to the first dose of administration, except for cancerous fever.
11. History of pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonia, drug-associated pneumonia or severely impaired lung function.
12. Inherited or acquired immunodeficiency disease, including but not limited to infection of HIV or active hepatitis (HBV DNA ≥ 1000 IU/ml or HCV RNA ≥ 1000 IU/ml).
13. Live vaccine administration within 4 weeks prior to the first dose of administration or probably during the study.
14. History of psychotropic substance abuse, alcohol abuse, or drug use.
15. Pregnancy or lactation
16. Exclusion from the study by the judgement of investigator, due to some factors that may lead to the forced termination of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2022-10-10 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Up to 2 years
  ORR is defined as the percentage of patients who have achieved complete response (CR) or partial response (PR), as measured by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria.

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to 2 years
  OS is defined as the time from first treatment to death, regardless of disease recurrence.
Progression-Free Survival (PFS) | Up to 2 years
  PFS is defined as the time from the first dose of administration to progression or death.
Disease control rate (DCR) | Up to 2 years
  DCR is defined as the percentage of patients who have achieved CR, PR or stable disease(SD), as measured by RECIST 1.1 criteria.
Incidence of Adverse Events (AE) | Up to 2 years
  The percentage of patients who suffer grade 3 or worse adverse events from the first dose of administration to last follow-up, assessed by the Common Terminology Criteria for Adverse Events (CTCAE) v5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Ming Kuang, PhD, Study Chair — First Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No